CLINICAL TRIAL: NCT04382209
Title: Evaluation of Ultrasound-Guided Erector Spinae Plane Block for Postoperative Analgesia in Adult Patients Undergoing Major Abdominal Surgery: A Prospective Randomized Controlled Clinical Trial
Brief Title: The Goal of This Study is to Evaluate the Effect of Ultrasound Guided Erector Spinae Plane Block on Postoperative Pain After Major Abdominal Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Bassem Mohammad Kamel EL-Ayashy, Assistant lecturer, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESPB for postoperative pain
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Pain
Keywords: Erector spinae plane block; Postoperative pain; Bupivacaine; Major abdominal surgeries; Meperidine; Intravenous patient controlled analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae plane block group (Active Comparator): Erector spinae plane block will be administrated to this group. An intravenous patient controlled analgesia device will be given to the patients postoperatively.
  Interventions: Procedure: Erector spinae plane block
- Control group (Sham Comparator): An intravenous patient controlled analgesia device will be given to the patients postoperatively
  Interventions: Device: Intravenous meperidine patient controlled analgesia device

INTERVENTIONS:
Procedure: Erector spinae plane block — The transducer was placed vertically 3cm lateral to the midline to visualize the muscles of the back, transverse process and the pleura in between the two transverse processes. Bilateral ultrasound guided erector spinae plane block with 20 mL of 0.375% bupivacaine each using an in-plane, cranial-to-caudad approach to contact the bony shadow of the transverse process (TP) with the tip deep to the fascial plane of the erector spinae muscle. The correct location of the needle tip was confirmed by injecting 0.5-1 cc of normal saline 0.9% and observing linear fluid spread lifting the erector spinae muscle off the tip of the TP.
  Arms: Erector Spinae plane block group
Device: Intravenous meperidine patient controlled analgesia device — Intravenous meperidine patient controlled analgesia device will be given to the patients postoperatively and 24 hour meperidine consumption will be recorded
  Arms: Control group

SUMMARY:
Aim of the work To evaluate the efficacy of ultrasound-guided erector spinae plane block for management of postoperative pain in patients undergoing major abdominal surgery under general anesthesia.

Hypothesis

* Null hypothesis: The investigators suppose that ultrasound-guided erector spinae plane block has no post-operative analgesic effect in patients undergoing major abdominal surgery.
* Alternative hypothesis: The investigators suppose that ultrasound-guided erector spinae plane block has post-operative analgesic effect in patients undergoing major abdominal surgery.

Study objectives

Primary Objective:

Comparison of opioid consumption in patients receiving erector spinae plane block in relation to control group.

Secondary Objective:

1. Evaluate the hemodynamics (blood pressure, heart rate) and respiratory rate in patients receiving erector spinae plane block during postoperative period at 0, 2, 4, 6, 8, 12,24 hours.
2. Assessment of numeric rating scale (NRS) in patients receiving erector spinae plane block during rest and movement during postoperative period at 0, 2, 4, 6, 8, 12,24 hours.

DETAILED DESCRIPTION:
Introduction:Thoracic epidural analgesia is still considered the gold standard for postoperative analgesia in abdominal surgery; however, concerns regarding side effects such as hypotension and motor blockade, as well as the risk of major complications such as epidural hematoma and abscess, have led some to question its role. Abdominal wall blocks such as the transversus abdominis plane (TAP) block have been proposed as alternatives; nevertheless they have their own limitations: dermatomal coverage is limited, catheter techniques are cumbersome to perform given the proximity to the surgical field, and a recent meta-analysis found the TAP block to be marginally effective in this context. The erector spinae plane (ESP) block is a novel paraspinal plane block first described for thoracic analgesia when performed at the T5 level, but more recently has also been shown to be effective in providing extensive somatic and visceral abdominal analgesia when performed at the T7-9 level.

Morphine administration is the cornerstone of pain therapy, but acute tolerance after opioid exposure has been described as early as the immediate postoperative period.Enhanced recovery after surgery, which involves implementation of evidence-based multimodal procedure- specific perioperative care pathways, has been shown to improve postoperative outcome and reduce length of hospital stay. One of the major elements of a successful program for enhanced recovery after surgery is the provision of optimal postoperative analgesia to facilitate ambulation and rehabilitation therapy.

An ideal multimodal analgesic technique would include local/regional analgesic techniques (i.e., neuraxial blocks [epidural and paravertebral analgesia], field blocks [e.g., transversus abdominis plane blocks and rectus sheath block], and surgical site infiltration) combined with acetaminophen and either a nonsteroidal antiinflammatory drug or a cyclooxygenase-2 selective inhibitor and also analgesic adjuncts such as single intraoperative dose dexamethasone.

The origin of pain from abdominal surgery is multifactorial, including a parietal (or somatic) component originating from the surgical incision and a visceral component originating from the peritoneum and the manipulation of the intra-abdominal structures. The somatic innervation of the anterior abdominal wall arises from the thoracolumbar spinal nerves (i.e., T6-L1).A recent cadaveric study assessing the course of anterior abdominal wall nerves found that there is extensive branching and communications between the abdominal nerves.The communications occur at several sites, including the intercostal plexus, anterolateral large branch communication, the transversus abdominis plane plexus that lies between the internal oblique and the transversus abdominis muscles (T9-L1 segmental nerves adjacent to the deep circumflex iliac artery), and the rectus sheath plexus that comprises all the segmental nerves (i.e., T9-L1) adjacent to the deep inferior epigastric artery. In most cases, these nerves also pierce the posterior surface of the rectus abdominis muscle.The muscular and cutaneous branches of these segmental nerves enter the muscle and finally terminate in the skin. The skin above the umbilicus is supplied by the cutaneous nerves derived from T6 to T9, the area around the umbilicus is innervated by T10, and the skin below the umbilicus is derived from T11, T12, and L1.

It is now evident that the peritoneum is a metabolically active organ and responds to surgical insult by manifesting a local and systemic immunologic and inflammatory response.The peritoneum consists of "silent nociceptors" that are activated by surgical injury and intraperitoneal inflammation and contribute to visceral pain. The neuro-immuno-humoral pain pathways involved in abdominal surgery include somatic and autonomic nerves such as the afferent fibers of the abdominal vagus nerve. Parasympathetic activation has been shown to influence perioperative outcome, as reduced vagal tone augments inflammation and increases gastrointestinal dysfunction.

Erector Spinae Plane Block (ESPB) - first recently described for the treatment of thoracic neuropathic pain, is a peri-paravertebral regional anesthesia technique that has since been reported as an effective technique for prevention of postoperative pain in various surgeries. In ESPB, local anesthetic is reported to be administered in to the interfascial plane between the transverse process of the vertebra and the erector spinae muscles, spreading to multiple paravertebral spaces. The ESP block was mentioned by the American society for regional anesthesia and pain medicine for pain management of rib fractures and described it as a paraspinal fascial plane block that involves injection of local anesthetic deep in the erector spinae muscle and superficial to the tips of the thoracic transverse processes. The site of injection is distant from the pleura, major blood vessels, and spinal cord; hence, performing the ESP block has relatively few contraindications. The ESP block is less difficult to perform relative to thoracic epidural anesthesia and thoracic paravertebral block. Case reports have reported that ESPB affects both the ventral and dorsal rami and leading to blockage of both visceral and somatic pain.

Ultrasound guided erector spinae (ESP) block is a regional anesthesia technique lead to analgesic effect on somatic and visceral pain by affecting the ventral rami and rami communicantes that include sympathetic nerve fibers, as local anesthetic spreads through the paravertebral space. When performed bilaterally it has been reported to be as effective as thoracic epidural analgesia.

In a study evaluating the effect of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy, they concluded that bilateral ultrasound guided ESPB leads to effective analgesia and a decrease in analgesia requirement in first 12 h in patients undergoing laparoscopic cholecystectomy, in which both somatic and visceral pain occurs .

Aim of the work :To evaluate the efficacy of ultrasound-guided erector spinae plane block for management of postoperative pain in patients undergoing major abdominal surgery under general anesthesia.

Hypothesis

* Null hypothesis: The investigators suppose that ultrasound-guided erector spinae plane block has no post-operative analgesic effect in patients undergoing major abdominal surgery.
* Alternative hypothesis: The investigators suppose that ultrasound-guided erector spinae plane block has post-operative analgesic effect in patients undergoing major abdominal surgery.

Study objectives

Primary Objective:

Comparison of opioid consumption in patients receiving erector spinae plane block in relation to control group.

Secondary Objective:

1. Evaluate the hemodynamics (blood pressure, heart rate) and respiratory rate in patients receiving erector spinae plane block during postoperative period at 0, 2, 4, 6, 8, 12,24 hours.
2. Assessment of numeric rating scale (NRS) in patients receiving erector spinae plane block during rest and movement during postoperative period at 0, 2, 4, 6, 8, 12,24 hours.

Study question:Is using ultrasound-guided erector spinae plane block effective in relieving postoperative pain in patients undergoing major abdominal surgery? Patients and methods After obtaining approval by the Institute Ethics Committee, and Written informed patient consent with an explanation regarding the purpose, methods, effects, and complications. The study will be performed on patients undergoing abdominal laparoscopic surgeries under general anesthesia. Patients will be randomly allocated to one of two equal groups.

Control group:

28 Patients will receive postoperative analgesia by intravenous patient controlled analgesia (IVPCA). Once pain is expressed by the patient or if the NRS is ≥ 4, patient will press a button and the IVPCA pump will programmed to deliver a bolus dose of 1 ml with 15 minutes lockout interval and no background infusion allowed. Each 1ml of IVPCA solution will contain 10 mg meperidine.

Erector Spinae plane block group:

28 Patients will have bilateral ultrasound guided erector spinae plane block with 20 mL of 0.375% bupivacaine each using an in-plane, cranial-to-caudad approach to contact the bony shadow of the transverse process with the tip deep to the fascial plane of the erector spinae muscle. The correct location of the needle tip is confirmed by injecting 0.5-1 cc of normal saline 0.9% and observing linear fluid spread lifting the erector spinae muscle off the tip of the TP.

Type of Study:

Prospective, randomized, comparative, double blinded clinical trial on an intention-to-treat basis.

Study setting:

Suez Canal University hospital elective surgical theaters.

Population and sample:

Patients who will undergo abdominal surgery in Suez Canal university hospitals in the elective surgical theaters .

Methods

Demographic data:

The patient's age, height, weight, ASA status, and duration of surgery will be recorded.

The ASA physical status classification system is a system for assessing the fitness of patients before surgery. The American Society of Anesthesiologists (ASA) adopted the five-category physical status classification system; a sixth category was later added. These are:

1. Healthy person.
2. Mild systemic disease.
3. Severe systemic disease.
4. Severe systemic disease that is a constant threat to life.
5. A moribund person who is not expected to survive without the operation.
6. A declared brain-dead person whose organs are being removed for donor purposes.

Medical history:

* Medical disorders as hypertension, diabetes, heart, chest, liver or kidney diseases.
* Past history of operations, hospitalization or blood transfusion
* Past anesthetic history with impact on previous airway problems during previous surgeries, hypersensitivity to anesthetic medications, any previous post-operative complications that could be attributed to anesthesia.
* Family history for specific anesthetic problems like malignant hyperthermia.

Physical examination:

* General examination & vital signs (heart rate, blood pressure, respiratory rate and temperature).
* Heart, chest and abdominal examinations.

Anesthetic assessment:

* Examination of the limbs for prediction of difficult cannulation.
* Airway assessment including:

A) Thyromental distance.

B) Mallampati score:

Class I: Soft palate, uvula, fauces, pillars visible. Class II: Soft palate, major part of uvula, fauces visible. Class III: Soft palate, base of uvula visible. Class IV: Only hard palate visible.

C) Neck and temporo-mandibular joint mobility. D) Examination of the airway mandible, tongue, palate, teeth and neck for any deformities that may interfere with airway management .

Laboratory investigations:

* Complete blood count.
* Prothrombin time and partial tissue thromboplastin time.
* Revision of metastatic workup.
* Electrolytes and random blood sugar.
* Liver and kidney function tests.

Technique:

Airway devices and anesthesia machine, ventilator, flowmeters and equipments will be checked promptly.

Patients will be monitored by Non-invasive blood pressure, pulse oximetry, and electrocardiogram prior to the induction of anesthesia.

Insertion of 20 G cannula in the upper limb. Pre-induction heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean arterial pressures (MAP) will be recorded as baseline values.

Induction of anesthesia for all participating patients is done with 2 μg/kg fentanyl, 1.5 - 2 mg/kg propofol. Endotracheal intubation will be facilitated by 0.15 mg/kg cis-atracurium. Anesthesia will be maintained by 1 - 1.5 minimum alveolar concentration (MAC) isoflurane in 50% oxygen/air mixture and 0.03 mg/kg cis-atracurium every 40 minutes.

Standard perioperative intravenous analgesia protocol included paracetamol 1 g, diclofenac sodium 75 mg. Analgesics will be supplemented by fentanyl 1μg/kg if the patient's hemodynamics (blood pressure & heart rate) increased after excluding light anesthesia.

The patients will be randomly assigned into 2 groups using a randomization-computer program.

All blocks were performed under sedation and analgesia, and before general anesthesia induction. Following routine monitoring and premedication the patients will be placed in the sitting position. ESPB was performed under ultrasonographic guidance using a linear 6- mega hertz (MHz) ultrasound probe (SonositeR, Inc. U.S.A). The linear ultrasound transducer was placed in a longitudinal parasagittal orientation 3 cm lateral to the T8 spinous process. The erector spinae muscles were identified superficial to the tip of the T8 transverse process. The patient's skin will be anesthetized with 3 ml of 2% lidocaine. A 21-gauge 10-cm needle was inserted using an in-plane superior-to-inferior approach. The tip of the needle was placed into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip was confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging. A total of 20 mL of 0.375% bupivacaine was injected.

Follow up vital signs (patient's heart rate, non-invasive blood pressure, oxygen saturation) during surgery every 15 minutes.

At the end of surgery, a reversal of the muscle relaxant is done using neostigmine (0.04 mg/kg) and atropine (0.01 mg/kg). After extubation, all patients will be transmitted to the post anesthesia care unit (PACU). Local anesthesia was not applied to wounds or nebulized intraperitoneally.

Postoperative analgesia will be given by intravenous patient controlled analgesia (IVPCA). The Numeric Rating Scale (NRS) was used to evaluate postoperative pain.

Numeric Rating Scale:

The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. It is considered a one dimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme ("no pain") to '10' representing the other pain extreme ("pain as bad as participants can imagine" or "worst pain imaginable"). Changes in NRS at rest and on movement were recorded at intervals.

Once pain is expressed by the patient or if the NRS is ≥ 4, patient will press a button and the IVPCA pump will programmed to deliver a bolus dose of 1 ml with 15 minutes lockout interval and no background infusion allowed. Each 1 ml of IVPCA solution will contain 10 mg meperidine.

All patients will be followed up and assessed at baseline and during surgery for vital signs (patients' heart rate, non-invasive arterial blood pressure, respiratory rate, and oxygen saturation). Post-operative they will be monitored for vital signs and the NRS score at 1 hour , 2 hours, 4 hours, 6 hours , 8 hours , 12 hours and 24 hours. Also, the time to first request of analgesia, and total meperidine consumption will be monitored in the 24 hours postoperative.

Statistical Analysis:

The statistical analysis will be performed using a Statistical Package for the Social Sciences SPSS® version 22 (SPSS Inc., Chicago, USA) for windows operating system.

Descriptive data will be expressed as mean and standard deviation (SD) for continuous variables, median and interquartile range for ordinal variables, and count and/or percentages (%) for discrete variables.

Independent-samples student T test will be used to analyze continuous variables between groups. One-way ANOVA will be used to analyze the parametric follow-up data within the same group. Discrete (categorical) variables will be analyzed using the Chi-square. The level of statistical significance is considered to be p<0.05.

Presentation of the statistical outcomes will be performed in a form of tables and graphs using the "Microsoft Office Excel® 2010" program.

Ethical Consideration:

1. The study procedures will be in accordance with the guidelines of Helsinki Declaration on human experimentation.
2. Written consent will be obtained from all patients after full explanation of hazards and benefits of the management procedures that will be performed for each patient before getting them involved in the study.
3. Bupivacaine (drug used in the study) is already approved by the Egyptian Drug Authority (EDA), marketed and used in clinical practice so; they have no additional harmful effects.
4. Patients have the right to refuse participation without affecting the medical care offered to them.
5. Patients have the right to withdraw from the study at any time without giving reasons, and this will not affect the medical care offered to them.
6. Confidentiality of all data and test results of all the study population will be preserved.
7. In case of failure of block , alternative plan will be ready and the patient will be excluded from study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 21 - 60 years
* Patients undergoing major abdominal surgery:

  * The indication for operation may be for benign or malignant disease.
  * Major surgery is defined as an operation of anticipated duration of more than one hour.

Exclusion Criteria:

* Patients with history of bleeding diathesis or on anticoagulant.
* Patients with relevant drug allergy.
* Patients with psychiatric illnesses, opioid dependence; alcohol or drug abuse that would interfere with perception and assessment of pain were excluded from the study.
* Compensated or decompensated myocardial insufficiency.
* Decreased renal function (serum creatinine <2.0 mg/dL).
* Infection of the skin at the site of needle puncture area

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours after surgery
  Meperidine consumptions for both group will be recorded

SECONDARY OUTCOMES:
Numeric rating scale (NRS) | 24 hours after surgery
  Numeric rating scale for pain will be used for pain evaluation during rest and movement . The scale is scored in a range of 0-10 with 0 representing no pain 10 representing the highest degree of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem M EL-Ayashy, Master Degree, Principal Investigator — Suez Canal University; Emad EL-Deen A Ibrahim, Doctor of Medicine, Study Director — Suez Canal University; Hamdy A Hendawy, Doctor of Medicine, Study Director — Suez Canal University
Locations (1):
- Suez Canal Teaching Hospital, Faculty of Medicine, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392